CLINICAL TRIAL: NCT03781947
Title: A Phase I, Open-label, Single Centre Study Investigating the PK, Safety and PD of a Single Dose of Teverelix TFA, a GnRH Antagonist, Via s.c. or i.m. Route of Administration in Healthy Male Volunteers
Brief Title: A Study of Parenterally-administered Teverelix TFA in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antev Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANT-1111-P01
Record Dates: First submitted 2018-11-19; First posted 2018-12-20 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This Phase I clinical study is an open-label, parallel-design, single-centre study to investigate the PK, safety and PD following subcutaneous and intramuscular administration of single doses of teverelix TFA in healthy male subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 90 mg s.c. (Experimental): A single s.c. injection of 90 mg teverelix TFA administered on Day 1
  Interventions: Drug: teverelix TFA
- 60 mg s.c. (Experimental): A single s.c. injection of 60 mg teverelix TFA administered on Day 1
  Interventions: Drug: teverelix TFA
- 90 mg i.m. (Experimental): A single i.m. injection of 90 mg teverelix TFA administered on Day 1
  Interventions: Drug: teverelix TFA
- 120 mg s.c. (Experimental): A single s.c. injection of 120 mg teverelix TFA administered on Day 1
  Interventions: Drug: teverelix TFA

INTERVENTIONS:
Drug: teverelix TFA — A single s.c. or i.m. injection of teverelix TFA administered on Day 1

SUMMARY:
A Phase I, open-label, single centre study investigating the pharmacokinetics, safety and pharmacodynamics of a single dose of teverelix TFA, a gonadotrophin releasing hormone antagonist, via subcutaneous or intramuscular route of administration in healthy male volunteers

DETAILED DESCRIPTION:
The primary objective of the study is:

• To characterise the pharmacokinetic (PK) profile of teverelix following single dose, subcutaneous (s.c.) and intramuscular (i.m.) administration of teverelix TFA in healthy male subjects

The secondary objectives of the study are:

* To assess the safety and tolerability of teverelix TFA after single s.c. and i.m. injections in healthy male subjects
* To evaluate pharmacodynamics (PD) effects of teverelix following single dose, s.c. and i.m. administration of teverelix TFA in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntarily agreement to participate in this study and sign an Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the screening procedures.
2. Males of any ethnic origin, between 40 to 70 years of age (inclusive) at the screening visit.
3. Healthy, determined by pre-study medical evaluation (medical history, vital signs, physical examination, standard 12-lead ECG and clinical laboratory evaluations).

   If a vital sign or ECG assessment is outside of the reference range at the screening visit or admission, the assessment may be repeated once to rule out any error.
4. Body mass index (BMI) between 20.0 and 34.9 kg/m2 (inclusive) at the screening visit and on admission.

Exclusion Criteria:

1. Clinically relevant history of cardiovascular, respiratory, hepatic, renal, pancreatic, gastrointestinal, metabolic, endocrine, neurological, dermatological, immunological, psychiatric or other diseases/disorders as determined by the Principal Investigator or designee, or evidence of such diseases/disorders during the screening period.
2. Any disorder or clinically relevant surgical history that would interfere with the absorption, distribution, metabolism or excretion of the study drug.
3. History of proneness to orthostatic dysregulation, fainting or blackouts.
4. History or physical evidence of chronic or clinically relevant acute infection.
5. Screening total testosterone <3.0 ng/mL (<10.4 nmol/L).
6. History of anaphylactoid reactions or hypersensitivity to teverelix or GnRH antagonists or any of the excipients of the products tested.
7. History of clinically relevant allergies or idiosyncrasies to medication or food.
8. History of regular alcohol consumption exceeding 21 units per week within 2 years of study entry.
9. History of illicit drug abuse within 2 years of study entry.
10. Any ECG abnormality of clinical relevance; ECG QT interval corrected for heart rate using Fridericia's correction (QTcF) > 450 ms at the screening visit.
11. Any clinically relevant findings in the laboratory tests, as judged by the Principal Investigator, at the screening visit and on admission; alanine aminotransferase (ALT) > 1.5 x the upper limit of normal (ULN) and/or aspartate aminotransferase (AST) > 1.5 x ULN and/or total bilirubin > 1.0 x ULN, as confirmed by subsequent repeat assessment, at the screening visit and on admission. If a laboratory assessment is outside of the reference range at the screening visit or admission, the assessment may be repeated once to rule out laboratory error.
12. An estimated glomerular filtration rate (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft Gault formula and normalised to an average surface area of 1.73m2, at the screening visit.
13. Positive results in any of the tests for hepatitis B surface antigen (HBsAg), total hepatitis B core antibody (HBcAb), hepatitis C antibody (anti-HCV) or human immunodeficiency virus (HIV) antibodies, at the screening visit.
14. Positive urine test for ethanol and/or drugs of abuse at the screening visit or admission.
15. Use of prescription, non-prescription and over-the-counter (OTC) medications (including vitamins or herbal remedies) within 2 weeks prior to dosing is prohibited.
16. Receiving an investigational product in a clinical trial within 3 months prior to the screening visit.
17. Donation of blood (> 500 mL) or blood products within 2 months (56 days) prior to the screening visit.
18. Unwilling to avoid consumption of coffee and caffeine-containing products within 48 hours prior to admission until discharge from the study centre, as well as from 48 hours before ambulatory visits.
19. Unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to admission until discharge from the study centre, as well as from 48 hours before ambulatory visits.
20. Unwilling to abstain from vigorous exercise from 72 hours prior to admission until discharge from the study centre, as well as from 72 hours before ambulatory visits.
21. Unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.
22. Subject is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
23. Subject has any concurrent condition that, in the opinion of the Principal Investigator, would make the subject unsuitable for participation in the clinical study.
24. Subject is an employee or the close relative of an employee of the Sponsor or the clinical research organisation (CRO) involved in the clinical study.
25. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male volunteers
Enrollment: 48 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 12 weeks
  Area under the concentration time-curve from time zero up to the last measurable concentration at time point t Area under the concentration time-curve from time zero up to the last measurable concentration at time point t Area under the concentration time-curve from time zero up to the last measurable concentration at time point t
AUC0-t1 | 12 weeks
  Area under the concentration time-curve from time zero up to concentration at time point t1 after which the concentrations start to rise again towards a second peak, t1 will be determined after review of the concentration-time profiles (immediate release component of total observed AUC)
AUCt1-t | 12 weeks
  Area under the concentration time-curve from time point t1 up to time point t (slow release component of total observed AUC)
AUC0-∞ | 12 weeks
  Area under the concentration time-curve from time zero up to infinity (∞)
Cmax | 12 weeks
  Maximum observed concentration after administration
Cmax,0-t1 | 12 weeks
  Maximum observed concentration after administration from zero up to time point t1
Cmax,t1-t | 12 weeks
  Maximum observed concentration after administration from time point t1 up to time point t
Tmax | 12 weeks
  Time to reach Cmax after dosing
Tmax,0-t1 | 12 weeks
  Time to reach Cmax,0-t1 after dosing
Tmax,t1-t | 12 weeks
  Time to reach Cmax,t1-t after dosing
λz | 12 weeks
  Apparent terminal rate constant
t½ | 12 weeks
  Apparent terminal plasma half-life

SECONDARY OUTCOMES:
Systemic tolerability - Incidence of Treatment-Emergent Adverse Events | 12 weeks
  Systemic tolerability assessed by incidence of treatment emergent AEs (TEAEs)
Local tolerability - Standardised Injection Site Reaction Scoring System (4-point) plus photography | 12 weeks
  The injections sites will be assessed (score 0 = none; 1 = mild; 2 = moderate; 3 = severe and undesirable) for signs of erythema, swelling, bruising, itching, pain and other signs of local reactions. Subjects will be monitored for duration of symptoms, sequelae and impact on activities of daily living (ADL). Photographs of all injection sites will be taken at all study visits post-administration
Cardiac assessments | 12 weeks
  The following 12-lead ECG parameters will be assessed: PR interval, QRS interval, RR interval, QT interval and QTc interval (QTcF)
24 hour Holter monitoring | Day -1 to Day 1
  Triplicate 10 second 12-lead ECGs will be extracted at time points prior to PK sampling times (Day 1) and matched timepoints (Day -1) in order to facilitate concentration-QTc effect modelling

OTHER OUTCOMES:
Testosterone (total) levels | 12 weeks
  Individual data listings of hormone level results will be presented for each subject
Luteinising Hormone (LH) levels | 12 weeks
  Individual data listings of hormone level results will be presented for each subject
Follicle Stimulating Hormone (FSH) levels | 12 weeks
  Individual data listings of hormone level results will be presented for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, MD, Principal Investigator — Parexel
Locations (1):
- PAREXEL International Early Phase Clinical Unit (EPCU), London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No